CLINICAL TRIAL: NCT03832595
Title: Kidney Coordinated Health Management Partnership
Acronym: Kidney-CHAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Vanderbilt University Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Manisha Jhamb, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19060280; R18DK118460 (NIH); 1R01DK116957-01A1 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-02-06 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Diseases
Keywords: electronic health record; population health management; patient education; medication therapy management; electronic consultation; randomized controlled trial; pragmatic trial
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial with randomization occurring at the Primary Care Physician practice level
Who Masked: Outcomes Assessor
Masking Description: outcomes are ascertained by data programmers who are blinded to study arm assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Patients in the usual care arm will continue to receive CKD care guided by their PCPs as per usual care practices (i.e., specialty consultation, pharmacotherapy, nurse education, etc. may be ordered by the PCP according to their usual practice).
  Interventions: Other: Usual Care
- Intervention Arm (Experimental): Patients will receive a care bundle
  Interventions: Other: EHR-based PHM

INTERVENTIONS:
Other: EHR-based PHM — An EHR in-basket message will be sent to the patient's PCP which identifies the patient's high-risk CKD status and indicates that the patient will receive:
  1. Nephrologist led electronic consultation: review of the patient's EHR with recommendations sent to the PCP every ~6 months,
  2. Medication therapy management: PharmD led telephonic medication therapy management with the patient every ~6 months,
  3. and Nurse led CKD patient education, every ~6-12 months
  unless the PCP opts the patient out of the interventions (by responding to the EHR in-basket message and providing an opt-out reason or requesting an office consultation with nephrology).
  Arms: Intervention Arm
Other: Usual Care — Patients in the usual care arm will continue to receive CKD care guided by their PCPs as per usual care practices (i.e., specialty consultation, pharmacotherapy, nurse education, etc. may be ordered by the PCP according to their usual practice).
  Arms: Usual care

SUMMARY:
As part of a 42-month pragmatic, cluster randomized trial in 1,650 primary care patients with high-risk Chronic Kidney Disease (CKD), the investigators will test the effectiveness of a multifaceted Electronic Health Record (EHR)-based Population Health Management (PHM) intervention that targets improvements in the delivery of evidence-based CKD care.

DETAILED DESCRIPTION:
To test the effectiveness of a multifaceted Electronic Health Record (EHR)-based Population Health Management (PHM) intervention to improve the delivery of evidence-based Chronic Kidney Disease (CKD) care in patients with high-risk CKD. Investigators will perform a 42-month pragmatic, cluster randomized (at the practice level) controlled trial in 1,650 patients with high-risk CKD (as defined by validated risk prediction models or by current estimated Glomerular Filtration Rate (eGFR) value or recent decline in eGFR values) managed by their Primary Care Physicians (PCPs) to determine whether EHR-based PHM improves key processes of care and clinical outcomes.

The investigators hypothesize that EHR-based PHM will improve hypertension control, use of renin angiotensin aldosterone system inhibitors (RAASi), and avoidance of renally contraindicated medications (Aim 1a-1c) and delay CKD progression (Aim 2).

Investigators will also characterize the acceptability and experience of Primary Care Physicians (PCPs) in the intervention arm of the CKD PHM study (Aim 3).

ELIGIBILITY:
Inclusion criteria for PCPs: presence of an ambulatory continuity clinic in the University of Pittsburgh Medical Center (UPMC) community medicine practice.

Inclusion criteria for patients:

1. age greater than or equal to 18, and less than or equal to 85
2. most recent eGFR less than 60 ml/min/yr
3. established care with UPMC PCP
4. high risk CKD based on validated external and internal risk prediction models or severe reduction in eGFR, or substantial loss in eGFR in prior 18 months.

Exclusion Criteria for PCPs: none

Exclusion Criteria for patients:

1. history of kidney transplant
2. receiving maintenance dialysis
3. recent (within 12 months) outpatient nephrology visit
4. baseline eGFR less than 15ml/min
5. expected survival less than 6 months or hospice enrollee (e.g., stage IV heart failure, metastatic cancer, oxygen dependent Chronic Obstructive Pulmonary Disease)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1596 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Abdel-Kader, MD, Principal Investigator — Vanderbilt University Medical Center; Manisha Jhamb, MD MPH, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jhamb M, Weltman MR, Yabes JG, Kamat S, Devaraj SM, Fischer GS, Rollman BL, Nolin TD, Abdel-Kader K. Electronic health record based population health management to optimize care in CKD: Design of the Kidney Coordinated HeAlth Management Partnership (K-CHAMP) trial. Contemp Clin Trials. 2023 Aug;131:107269. doi: 10.1016/j.cct.2023.107269. Epub 2023 Jun 20. PMID 37348600
- [Derived] Jhamb M, Weltman MR, Devaraj SM, Lavenburg LU, Han Z, Alghwiri AA, Fischer GS, Rollman BL, Nolin TD, Yabes JG. Electronic Health Record Population Health Management for Chronic Kidney Disease Care: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2024 Jul 1;184(7):737-747. doi: 10.1001/jamainternmed.2024.0708. PMID 38619824
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37348600/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18,157 participants from 101 practices underwent initial screening. Out of these 1,803 from 9 practices were eligible at initial screening, which included 874 (from 50 practices) in control arm, and 929 (from 4 practices) in intervention arm.
  Patients who had confirmed eligibility after initial screening and had a PCP appointment within 1 year of eligibility screening were enrolled. In intervention group, patients or PCPs who opted-out at this stage were not enrolled
Units Other Than Participants: Primary care practices
Groups:
- Intervention Arm: Patients will receive a care bundle
  EHR-based PHM: An EHR in-basket message will be sent to the patient's PCP which identifies the patient's high-risk CKD status and indicates that the patient will receive:
  1. Nephrologist led electronic consultation: review of the patient's EHR with recommendations sent to the PCP every ~6 months,
  2. Medication therapy management: PharmD led telephonic medication therapy management with the patient every ~6 months,
  3. and Nurse led CKD patient education, every ~6-12 months
  unless the PCP opts the patient out of the interventions (by responding to the EHR in-basket message and providing an opt-out reason or requesting an office consultation with nephrology).
Period: Overall Study
Arm/Group | Intervention Arm | Usual Care
Started (These are patients who were eligible at initial screening) | 754; 48 Primary care practices | 842; 50 Primary care practices
Completed | 575; 48 Primary care practices | 711; 50 Primary care practices
Not Completed | 179; 0 Primary care practices | 131; 0 Primary care practices
Not completed — Death | 142 | 130
Not completed — Medical management without dialysis | 37 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Primary care practice
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Usual Care | Total
Number analyzed (Participants) | 754 | 842 | 1596
Number analyzed (Primary care practice) | 48 | 50 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.8 (9.1) | 73.4 (8.8) | 73.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 409 | 519 | 928
  Male | 345 | 323 | 668
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 748 | 831 | 1579
  Unknown or Not Reported | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 51 | 76 | 127
  White | 696 | 753 | 1449
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 754 | 842 | 1596
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 131.1 (16.6) | 131.6 (17.2) | 131.4 (16.9)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 73.9 (10.4) | 74.4 (10.8) | 74.1 (10.6)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.7 (0.4) | 1.7 (0.4) | 1.7 (0.4)
eGFR CKD-EPI [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 37.1 (7.9) | 36.6 (7.9) | 36.8 (7.9)
Urine Albumin-creatinine ratio [Median (Inter-Quartile Range); unit: UACR mg/g] | 86.0 [16.3 to 434.0] | 84.6 [14.0 to 410.3] | 85.0 [15.1 to 421.5]

OUTCOME MEASURES:

1. Primary Outcome: Renal Failure Event Defined as Greater Than or Equal to 40% Decline in Estimated Glomerular Filtration Rate (eGFR) or Occurrence of End Stage Renal Disease (ESRD)
Description: The outcome measure is occurrence of renal failure event and is defined as a greater than or equal to 40% decline in eGFR or occurrence of End Stage Renal Disease. The 40% decline in renal failure is a well accepted endpoint for renal failure in clinical trials and is approved by the FDA.
  eGFR decline will be adjudicated based on the baseline creatinine and eGFR determined from the CKD-epidemiology (CKD-EPI) equation and measured routinely in clinical practice. All eGFR values within 6-month windows will be averaged to account for ascertainment bias, and analyzed using discrete-time survival approach using generalized linear mixed model.
  ESRD will be defined as an eGFR less than or equal to 10ml/min, or starting of renal replacement therapy (dialysis or kidney transplant)
Time Frame: Time to event analysis - until primary outcome or a competing event (death, medication management without dialysis, being moved to hospice care) was achieved or until the end of intervention period (max 39 months). Cumulative % at 24 months reported
Measure: Number (95% Confidence Interval); unit: percent
Units Other Than Participants: Primary care practice
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 754 | 842
Number analyzed (Primary care practice) | 48 | 50
percent | 9.7 [6.6 to 12.7] | 10.9 [7.7 to 14.1]
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care; Test type: Equivalence — We determined that 1,653 patients provide 80% power to detect a hazard ratio of 0.64, or a 5% absolute risk reduction in intervention arm, assuming a primary end-point rate of 15% in the usual care group at 24 months, 20% loss to follow-up, α = 0.05, and within-practice intra-class correlation of 0.01; p = 0.82, Mixed Models Analysis; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.67 to 1.38]

2. Secondary Outcome: Hypertension (HTN) Control Outcome
Description: HTN control is defined as achieved BP<140/90mmHg. Outpatient, sitting Blood Pressure (BP) values measured during each outpatient encounter and recorded in the EHR. All BPs within a 6-month window are averaged to account for ascertainment bias and then analyzed using generalized linear mixed model for average BP as binary outcome. Result is reported as log-odds per month slope for each arm. Higher log-odds indicates higher rate of BP control
Time Frame: Time to event analysis - until primary outcome or a competing event (death, medication management without dialysis, being moved to hospice care) was achieved or until the end of intervention period (max 39 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: log-odds per month slope
Units Other Than Participants: Primary care practices
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 754 | 842
Number analyzed (Primary care practices) | 48 | 50
log-odds per month slope | 0.011 [-0.002 to 0.024] | 0.0005 [-0.012 to 0.013]
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care; Test type: Equivalence — α = 0.05; Slope difference = 0.011, 95% CI 2-sided [-0.008 to 0.029]

3. Secondary Outcome: Renin-Angiotensin-Aldosterone System Inhibitors (RAASi) Exposure Days Per Year
Description: Will be determined by active use of an Angiotensin-Converting Enzyme inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) based on the EHR medication list at each outpatient encounter (cumulative person-time exposure during the study). Reported as exposure days per year rate for each arm
Time Frame: Time to event analysis- Follow-up duration until primary outcome or a competing event (death, medication management without dialysis, being moved to hospice care) was achieved or until the end of intervention period (max 39 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: exposure days per year
Units Other Than Participants: Primary care practice
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 754 | 842
Number analyzed (Primary care practice) | 48 | 50
exposure days per year | 196.8 [174.9 to 219.0] | 163.1 [146.3 to 179.9]
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care; Test type: Equivalence — α = 0.05; Rate ratio = 1.21, 95% CI 2-sided [1.02 to 1.43]

4. Secondary Outcome: Medication Safety: Non-Steroidal Anti-inflammatory Drugs (NSAIDS) Exposure Days Per Year
Description: Investigators will examine the rates of use of several high-risk medications that can be associated with adverse outcomes in progressive CKD. Medication exposure will be determined by presence of the specified medication on the patient's EHR medication list at each outpatient encounter (cumulative person-time exposure during the study). Reported as exposure days per year rate for each arm NSAIDS use will be examined for all study patients
Time Frame: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: exposure days per year
Units Other Than Participants: Primary care practice
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 754 | 842
Number analyzed (Primary care practice) | 48 | 50
exposure days per year | 5.3 [2.6 to 8.0] | 6.7 [3.7 to 9.7]
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care; Test type: Equivalence — α = 0.05; Rate ratio = 0.80, 95% CI 2-sided [0.51 to 1.25]

5. Secondary Outcome: Medication Safety: Glyburide Exposure Days Per Year
Description: Investigators will examine the rates of use of several high-risk medications that can be associated with adverse outcomes in progressive CKD. Medication exposure will be determined by presence of the specified medication on the patient's EHR medication list at each outpatient encounter (cumulative person-time exposure during the study). Reported as Exposure days per year rate for each arm
  Glyburide use will be examined for all study patients with diabetes at baseline
Time Frame: Time to event analysis - Follow-up duration until primary outcome or a competing event (death, medication management without dialysis, being moved to hospice care) was achieved or until the end of intervention period(max 39 months)
Measure: Least Squares Mean (95% Confidence Interval); unit: exposure days per year
Units Other Than Participants: Primary care practice
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 467 | 534
Number analyzed (Primary care practice) | 48 | 50
exposure days per year | 2.4 [-3.7 to 8.5] | 2.0 [-1.6 to 5.7]
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care; Test type: Equivalence — α = 0.05; Rate ratio = 1.18, 95% CI 2-sided [0.03 to 53.78]

6. Secondary Outcome: Medication Safety: Metformin Exposure Days Per Year
Description: Investigators will examine the rates of use of several high-risk medications that can be associated with adverse outcomes in progressive CKD. Medication exposure will be determined by presence of the specified medication on the patient's EHR medication list at each outpatient encounter (cumulative person-time exposure during the study). Reported as Exposure days per year rate for each arm Use of metformin will be examined for all study patients with diabetes at baseline and eGFR less than 30
Time Frame: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: exposure days per year
Units Other Than Participants: Primary care practice
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 70 | 97
Number analyzed (Primary care practice) | 48 | 50
exposure days per year | 17.8 [-6.5 to 42.2] | 16.0 [-1.7 to 33.6]
Statistical Analysis 1: Comparison: Intervention Arm vs Usual Care; Test type: Equivalence — α = 0.05; Rate ratio = 1.12, 95% CI 2-sided [0.12 to 9.96]

7. Secondary Outcome: Medication Safety: Gemfibrozil Exposure Days
Description: We will examine the rate of use of gemfibrozil among those with eGFR<30 at baseline
Time Frame: Time to event analysis - Follow up duration until primary outcome or a competing event was achieved or until end of intervention period (max 39 months)
Population: Although Gemfibrozil was a pre-specified secondary outcome, it was excluded from analyses since among those with eGFR<30 at baseline, active use was found only in 1 patient control arm) and there is no statistically meaningful way of analyzing this
Units Other Than Participants: Primary care practice
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 0 | 0
Number analyzed (Primary care practice) | 0 | 0

8. Other Pre Specified Outcome: Subgroup Analysis: Use of Renin-Angiotensin-Aldosterone System Inhibitors (RAASi) (Outcome 3) in Participants With UACR ≥300 mg/g
Description: Outcome 3 will be repeated in the subgroup of participants receiving RAASi who have macroalbuminuria, RAASi use will be determined by active use of an Angiotensin-Converting Enzyme inhibitor (ACEi) or Angiotensin Receptor Blocker (ARB) based on the EHR medication list at each outpatient encounter (cumulative person-time exposure during the study).
Time Frame: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: medication exposure days per year
Arm/Group | Usual Care | Intervention Arm
Number analyzed (Participants) | 233 | 226
medication exposure days per year | 177.5 [146.2 to 208.8] | 222.5 [182.9 to 262.1]

9. Other Pre Specified Outcome: Hypertension (HTN) Control for Achieved BP <130/80 mm Hg
Description: HTN control is defined as achieved BP<130/80mmHg. Outpatient, sitting Blood Pressure (BP) values measured during each outpatient encounter and recorded in the EHR. All BPs within a 6-month window are averaged to account for ascertainment bias and then analyzed using generalized linear mixed model for average BP as binary outcome. Result is reported as log-odds per month slope for each arm. Higher log-odds indicates higher rate of BP control
Time Frame: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: log-odds per month slope
Arm/Group | Intervention Arm | Usual Care
Number analyzed (Participants) | 754 | 842
log-odds per month slope | 0.086 [0.073 to 0.100] | 0.079 [0.066 to 0.092]

ADVERSE EVENTS:
Time Frame: Over the entire study follow-up period, median follow-up 17 months
Arm/Group | Intervention Arm | Usual Care
All-Cause Mortality (participants affected / at risk) | 142/754 | 130/842
Serious Adverse Events (participants affected / at risk) | 18/754 | 21/842
Other Adverse Events (participants affected / at risk) | 59/754 | 77/842
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=754) | Usual Care (N=842)
Severe Hyperkalemia (Renal and urinary disorders) | 18 (23) | 21 (28) — Electrolytes
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=754) | Usual Care (N=842)
Moderate hyperkalemia (Serum potassium 5.5 - 6 meQ/L) (Renal and urinary disorders) | 59 (87) | 77 (107) — Electrolytes

LIMITATIONS AND CAVEATS:
Lower duration of follow-up period due to COVID-19 pandemic related delays

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03832595/Prot_SAP_000.pdf